CLINICAL TRIAL: NCT04863313
Title: Evaluation of the Effect of the Administration of a Probiotic Formulation on Glycemic Control, Insulin Resistance and the Composition of the Microbiota in Subjects With Prediabetes
Brief Title: Effect of a Probiotic on the Glycemic Profile and the Fecal Microbiota of Prediabetic Subjects (PREDIABETCARE)
Acronym: PREDIABETCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: GENBIOMA Aplicaciones SL (Unknown); Gobierno de Navarra/FEDER (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PREDIABETCARE
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2022-02

CONDITIONS: PreDiabetes; Overweight and Obesity
Keywords: Prediabetes; Obesity and overweight; Glycated hemoglobin; Blood glucose; Fecal microbiota; Probiotic
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving the probiotic capsules (Experimental): Experimental group will consume one probiotic capsule every day during 12 weeks at breakfast.
  Interventions: Dietary Supplement: Probiotic
- Group receiving the placebo capsules (Placebo Comparator): Placebo group will consume one placebo capsule every day during 12 weeks at breakfast.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Experimental group will consume one probiotic capsule every day during 12 weeks at breakfast.
  Arms: Group receiving the probiotic capsules
Dietary Supplement: Placebo — Placebo group will consume one placebo capsule every day during 12 weeks at breakfast.
  Arms: Group receiving the placebo capsules

SUMMARY:
According to the data from the Di@bet.es study, which is part of the National Diabetes Strategy, the prevalence of type 2 diabetes among Spanish population is 13.8%. Diabetic patients suffer from several short and long term complications, which are related to a significant worsen of quality of life and a substantial increase in death rate.

In this sense, it is important to prevent the development of Type 2 diabetes. Therefore, it is of high relevance to identify and to treat prediabetic subjects prior to the development of the disease. Many strategies have been implemented to reverse this situation, such as changes in diet and lifestyle, among others. However, it is hard to achieve changes in lifestyle and despite the use of some drugs in this phase of the disease, the problem continues growing.

For this reason, new strategies to combat the development of type 2 diabetes are been investigated, such as the use of probiotic formulations. However, at the moment, few studies evidence the effect of probiotics on glycemic regulation. Therefore, an interesting opportunity arises according to the potential ability of probiotic formulation for the control of prediabetes.

Considering this background, the main objective of this research is to assess the effect of a new probiotic formulation on glycemic control, insulin resistance and the composition of the fecal microbiota in prediabetic subjects.

DETAILED DESCRIPTION:
This study is designed as a 12-week, double-blind, randomised, placebo-controlled parallel study. It is focused on prediabetic overweight / obese men and women between 18 and 70 years old.

All participants attend the Nutrition Intervention Unit of the Center for Nutrition Research in the University of Navarra for the screening visit and 4 more times during the intervention (week 1, 4, 8 and 12 of study).

* Screening visit: evaluation of the inclusion criteria.

Volunteers who meet the inclusion criteria are provided with a stool collection kit and a 72 h food record questionnaire. Moreover, they are randomly assigned to one of the two intervention groups:

Control group: placebo supplemented; Experimental group: probiotic supplemented.

* Clinical investigation day 1 (day 1): The volunteer attend the Nutrition Intervention Unit in fasting state. Each volunteer is asked to provide the stool sample and the 72-hour food record questionnaire. Then, anthropometric, body composition and blood pressure measurements are taken and the gastrointestinal symptoms questionnaire is completed. After that, volunteer is provided with the capsules of the study for one month. Finally, fasting blood samples are collected and then an oral glucose tolerance test is carried out and blood samples are taken at 30, 60, 90 and 120 minutes after the ingestion of the glucose solution.
* Clinical investigation day 2 (week 4): The volunteer attend the Nutrition Intervention Unit in fasting state. The gastrointestinal symptoms questionnaire is completed and the adherence to the study and to the capsule consumption is assessed. After the measurement of anthropometric, body composition and blood pressure a blood sample is collected. Finally, volunteer is provided with capsules for the next month.
* Clinical investigation day 3 (week 8): The volunteer attend the Nutrition Intervention Unit in fasting state. The gastrointestinal symptoms questionnaire is completed and the adherence to the study and to the capsule consumption are assessed. After the measurement of anthropometric, body composition and blood pressure, a blood sample is collected. Finally, the stool collection kit, 72h food record questionnaire and capsules for one month are given to the volunteer.
* Clinical investigation day 4 (week 12): The volunteer attend the Nutrition Intervention Unit in fasting state. Each volunteer is asked to provide the stool sample and the 72-hour food record questionnaire. Then, anthropometric, body composition and blood pressure measurements are taken and the gastrointestinal symptoms questionnaire are completed. Finally, fasting blood samples are collected and then an oral glucose tolerance test is carried out and blood samples are taken at 30, 60, 90 and 120 minutes after the ingestion of the glucose solution.

One month later, the online version of the gastrointestinal symptoms questionnaire is send to each volunteer in order to asess any gastrointestinal symptom after stopping capsule consumption.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 70 years.
* Prediabetic subjects: glycosylated hemoglobin (HbA1c) between 5.7% and 6.4%.
* Body Mass Index (BMI) between 25 and 39.9 kg / m2.
* No weight changes (± 3 kg) during the last 3 months.
* The subjects must be in general physical and psychological conditions in accordance with the objective of the study.
* Subjects must be able to understand and sign the informed consent.

Exclusion Criteria:

* To be in continuous pharmacological / hormonal treatment, especially those that could affect blood glucose concentration.
* Suffering from a chronic metabolic disease, or from a systemic intestinal, liver or kidney disease: type 1 or 2 diabetes, severe dyslipidemia, uncontrolled thyroid function disorders, cirrhosis, inflammatory bowel disease, etc.
* Subjects suffering from severe hyperlipidemia, severe hypertension or hypothyroidism without treatment or treated for less than 3 months.
* Presence of relevant functional or structural abnormalities of the digestive system, such as malformations, angiodysplasia, active peptic ulcers, chronic inflammatory diseases or malabsorption.
* Subjects who have undergone gastrointestinal surgery with permanent sequelae (for example, gastroduodenostomy).
* Chronic treatment with stomach protectors.
* Subjects suffering from some type of cancer or being in treatment for it or with a period less than 5 years since its eradication.
* Presence of some type of mental impairment such as depressive pathology, anxiety or untreated bipolar disorder. They will be able to participate if they have stable treatment for at least 3 months prior to the begining of the trial.
* Allergy or intolerance to any food or food group that is likely to manifest during the study.
* Be on a special diet (Atkins, vegetarian, etc.) during the 3 months prior to the start of the study.
* Weight variations (± 3 kg) during the last 3 months.
* Suffering from eating disorders or eating restrictive behaviors (score on the EAT-26 questionnaire equal or greater than 20).
* Subjects who have undergone surgical treatment for obesity.
* Being pregnant or breastfeeding.
* Abuse of alcohol (more than 14 units in women and 20 units in men) and / or drugs.
* Show poor collaboration or, in the opinion of the investigator, have difficulties in following the study procedures.
* Take some type of nutritional supplementation that can affect blood glucose and / or microbiota. If they take it, in order to be included in the study, they will have to stop the supplement, with a washout period of at least 14 days before starting the study.
* People who are positive for Covid-19 will not be able to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Change of blood glycated hemoglobin (HbA1c) concentration from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Fasting blood glycated hemoglobin (HbA1c) concentration will be reported in % and in mmol/mol.

SECONDARY OUTCOMES:
Change of metagenomic analysis of intestinal microbiota composition from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Measured by analyzing the variable regions V3-V4 of the prokaryotic 16S rRNA (ribosomal ribonucleic acid) gene sequences.
Change of fasting blood glucose concentration from baseline to week 4. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Blood glucose concentration will be analyzed after an overnight fast.
Change of fasting blood glucose concentration from baseline to week 8. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Blood glucose concentration will be analyzed after and overnight fast.
Change of fasting blood glucose concentration from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Blood glucose concentration will be analyzed after an overnight fast.
Oral glucose tolerance test | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Blood glucose will be reported in mg/dl at 30, 60, 90 and 120 minutes as part of the oral glucose tolerance test
Change in the Area under the curve for glucose from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Area under the curve will be calculated using glucose levels after oral glucose tolerance test.
Change of fasting blood insulin concentration from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Blood insulin concentration will be analyzed after an overnight fast by ELISA kit.
Change of HOMA index from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  HOMA index will be calculated to analyze insulin resistance
Change of blood glucagon like peptide-1 (GLP-1) concentration from baseline to week 12. | The Time Frame contains two time points: day 1 (at baseline) compared to day 4 (after 12 weeks of intervention).
  Blood GLP-1 concentration will be analyzed after an overnight fast with ELSA kit.
Change of Blood peptide-C concentration from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Blood peptide-C concentration will be analyzed after and overnight fast.
Change of gastrointestinal symptoms from baseline to week 4. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Gastrointestinal symptoms will be analyzed by a gastrointestinal symptom questionnaire.
Change of gastrointestinal symptoms from baseline to week 8. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Gastrointestinal symptoms will be analyzed by a gastrointestinal symptom questionnaire.
Change of gastrointestinal symptoms from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Gastrointestinal symptoms will be analyzed by a gastrointestinal symptom questionnaire.
Change of blood ALT concentration from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Blood ALT concentration will be measured after an overnight fast.
Change of blood AST concentration from baseline to week 12. | The Time Frame contains two time points: day 1 (at baseline) compared to day 4 (after 12 weeks of intervention).
  Blood AST concentration will be measured after an overnight fast.
Change of blood total cholesterol concentratio from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Blood total cholesterol concentration will be analyzed after an overnight fast.
Change of blood HDL cholesterol concentration from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Blood HDL cholesterol concentration will be analyzed after an overnight fast.
Change of blood LDL cholesterol concentration from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Blood LDL concentration will be reported in mg/dl by Friedewald equation.
Change of blood triglyceride concentration from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Blood triglyceride concentration will be analyzed after an overnight fast.
Change of hemogram from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Blood hemogram
Change of weight from baseline to week 4. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Weight of participants in fasting condition will be analyzed by bioimpedance and reported in kg.
Change of weight from baseline to week 8. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Weight of participants in fasting condition will be analyzed by bioimpedance and reported in kg.
Change of weight from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Weight of participants in fasting condition will be analyzed by bioimpedance and reported in kg.
Change of body mass index from baseline to week 4. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Weight and height will be combined to report BMI in kg/m^2.
Change of body mass index from baseline to week 8. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Weight and height will be combined to report BMI in kg/m^2.
Change of body mass index from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Weight and height will be combined to report BMI in kg/m^2.
Change of waist circumference from baseline to week 4. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Waist circumference will be measured with a measuring tape and will be reported in cm.
Change of waist circumference from baseline to week 8. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Waist circumference will be measured with a measuring tape and will be reported in cm.
Change of waist circumference from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Waist circumference will be measured with a measuring tape and will be reported in cm.
Change of hip circumference from baseline to week 4. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Hip circumference will be measured with a measuring tape and will be reported in cm.
Change of hip circumference from baseline to week 8. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Hip circumference will be measured with a measuring tape and will be reported in cm.
Change of hip circumference from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Hip circumference will be measured with a measuring tape and will be reported in cm.
Change of body composition (fat mass, lean mass and water content) from baseline to week 4. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Body composition will be analyzed at fasting state by bioimpedance.
Change of body composition (fat mass, lean mass and water content) from baseline to week 8. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Body composition will be analyzed at fasting state by bioimpedance.
Change of body composition (fat mass, lean mass and water content) from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Body composition will be analyzed at fasting state by bioimpedance.
Change of systolic blood pressure from baseline to week 4. | The Time Frame contains two time points: day 1 (at baseline) compared to day 2 (after 4 weeks of intervention).
  Fasting systolic blood pressure will be measured by a tensiometer and reported in mmHg.
Change of systolic blood pressure from baseline to week 8. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Fasting systolic blood pressure will be measured by a tensiometer and reported in mmHg.
Change of systolic blood pressure from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Fasting systolic blood pressure will be measured by a tensiometer and reported in mmHg.
Change of dyastolic blood pressure from baseline to week 4. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Fasting dyastolic blood pressure will be measured by a tensiometer and reported in mmHg.
Change of dyastolic blood pressure from baseline to week 8. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Fasting dyastolic blood pressure will be measured by a tensiometer and reported in mmHg.
Change of dyastolic blood pressure from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Fasting dyastolic blood pressure will be measured by a tensiometer and reported in mmHg.
Change of heart rate from baseline to week 4. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Fasting heart rate will be measured by a tensiometer.
Change of heart rate from baseline to week 8. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Fasting heart rate will be measured by a tensiometer.
Change of heart rate from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Fasting heart rate will be measured by a tensiometer.
Change of physical activity from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Physical Activity will be analyzed by the International Physical Activity Questionnaire.
Change on food intake from baseline to week 12. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Energy and macronutrient intake will be analyzed by a 72h foor record questionnaire.
Adherence to the intervention at week 4. | Clinical investigation day 2 (week 4).
  Adherence to the intervention will be assessed by a capsule intake diary.
Adherence to the intervention at week 8. | Clinical investigation day 3 (week 8).
  Adherence to the intervention will be assessed by a capsule intake diary.
Adherence to the intervention at week 12. | Clinical investigation day 4 (week 12).
  Adherence to the intervention will be assessed by a capsule intake diary.

CONTACTS AND LOCATIONS:
Overall Officials: María Jesús Moreno Aliaga, PhD, Principal Investigator — University of Navarra; Carlos González Navarro, PhD, Study Director — University of Navarra; Pedro González Muniesa, PhD, Study Chair — University of Navarra; Idoia Ibero Baraibar, PhD, Study Chair — University of Navarra
Locations (1):
- Center for Nutrition Research. University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No